CLINICAL TRIAL: NCT01291888
Title: Efficacy and Tolerability of Nebivolol Versus Sustained Release Metoprolol Succinate in Patients With Chronic Kidney Disease: A Single-center Randomized Trial.
Brief Title: Nebivolol Versus Sustained Release Metoprolol Succinate in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Rajiv Saran, MBBS, MD, MS, MRCP, University of Michigan
Other Study IDs: HUM00034784
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A total of 30 ml blood (CBC with differential and platelets-3ml, comprehensive panel-5-7ml, biomarkers-20ml) will be drawn by venipuncture typically from the antecubital vein at baseline visit (30ml), and week 6-study midpoint (30ml) and end of study (30ml). At the screening visit only 10ml blood will be required (CBC and Comprehensive Panel).
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators postulate that nebivolol will be more effective than an equivalent dose of a comparative BB, specifically sustained release metoprolol succinate, in improving the availability of NO, lowering blood pressure, and reducing albuminuria with implications for slowing progression of CKD and cardiovascular protection in this high risk population.

The objective of this proposal is to conduct a randomized pilot clinical trial to determine the relative efficacy and tolerability of nebivolol versus sustained release metoprolol succinate in improving blood pressure in patients with CKD and albuminuria. The primary endpoint would be a decrease in asymmetric dimethyl arginine (ADMA). Secondary endpoints would include a reduction in blood pressure, urinary F2-isoprostanes and albuminuria.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) are at an increased risk of mortality related to cardiovascular (CV) disease compared with the general population. Furthermore, a reduced glomerular filtration rate (GFR), defined as < 60 ml/min/1.73m², has been shown to be associated with increased risk of hospitalization, death and cardiovascular events independent of other known cardiovascular risk factors.

Albuminuria, a marker of endothelial dysfunction or kidney damage, or both, frequently accompanies a reduction in GFR during the development of CKD, and is a well-recognized risk factor for kidney disease progression. Importantly, the presence of albuminuria has also been shown to be a powerful predictor of CV mortality independent of other risk factors.

Endothelial dysfunction has been implicated in the pathophysiology of progressive renal disease and may be a link between CKD and CV mortality. Levels of asymmetric dimethyl arginine (ADMA), a competitive inhibitor of nitric oxide synthase, are elevated in patients with CKD. Elevated levels of ADMA have been shown to correlate with the presence of endothelial dysfunction and to predict mortality in patients with CKD. In addition, ADMA has been shown to be associated with progression of non-diabetic kidney disease and lowering ADMA levels could potentially prevent progressive renal impairment.

Oxidative stress also plays a fundamental role in the development of endothelial function and cardiovascular disease. While markers of oxidative stress are notoriously difficult to measure, F2- isoprostanes are considered to be reliable biomarkers of in vivo lipid peroxidation. F2-isoprostanes are a family of prostaglandin F2 isomers produced by free radical peroxidation of arachidonic acid and have been used as end points in clinical studies of anti-oxidant therapies.

Blood pressure control is an important factor in predicting CV mortality. However, in patients with CKD, blood pressure is frequently difficult to control. Angiotensin converting enzyme inhibitors (ACEIs), and angiotensin receptor blockers (ARBs) with or without diuretics, are the antihypertensive agents of choice in patients with CKD. More recently, the combination of an ACEI and a dihydropyridine calcium channel blocker (CCB) have been shown to be more effective than an ACEI and a thiazide diuretic in controlling blood pressure in patients with essential hypertension including those with CKD or diabetes mellitus. However, even with this combination of medications, blood pressure control in patients with CKD is often difficult to achieve. The effect of beta adrenergic blocking agents (BB) on lowering blood pressure has not been extensively investigated in patients with CKD. A randomized control trial in hemodialysis patients from Italy showed that there was a higher two-year survival in those receiving carvedilol. Beta blockers are not routinely used to lower blood pressure in patients with CKD due to the possibility that these medications may have a deleterious effect on insulin resistance, although this theory has been disproved in a large clinical trial. A recent review points out that beta blockers are underused in patients with CKD although they offer many potential benefits in this patient population. This is not surprising, as sympathetic overactivity is an important contributor to cardiovascular disease and propensity to sudden death in patients with CKD. However, despite the potential benefits of BBs in patients with CKD their use remains limited because of the potential for inducing a relatively high rate of adverse effects and the lack of data in regard to their effectiveness in patients with CKD.

The recent availability of the third generation beta blocker nebivolol, known to improve the availability of nitric oxide by reducing ADMA levels, thereby improving endothelial function, provides an opportunity to more effectively control blood pressure, prevent the progression of CKD, and also the occurrence of CV events. A reduction in the bioavailability of nitric oxide (NO) has been shown to play a significant role in both endothelial dysfunction and hypertension. Therefore, increasing the availability of nitric oxide can potentially be very beneficial. In a comparative study in patients with diabetes mellitus a trial of nebivolol versus metoprolol showed that metoprolol raised ADMA levels, suggesting a worsening of endothelial function, whereas nebivolol did not have this effect. Thus, nebivolol would appear to have a major advantage over other BBs in patients CKD due to diabetes mellitus or hypertension although this has not yet been systematically studied.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old and < 85 years old
* Willing and able to comply with all study procedures
* Blood pressure on standard antihypertensive therapy, which may include: a diuretic, ACE-I, ARB, CCB, and/or an alpha adrenergic antagonist, and a blood pressure ≤ 180 mm Hg systolic and ≥ 130 mm Hg systolic. The blood pressure will be taken after a period of 15 minutes of resting in the sitting posture
* Clinically stable patients with CKD (GFR 20-60 ml/min/1.73 m²) by the abbreviated MDRD equation and with a rate of decline of GFR no greater than 1 ml/min/1.73 m² per month over the prior three months and with albuminuria (urine albumin:creatinine ratio) in a spot urine sample of between 100-3000 mcg/g of creatinine). Albumin excretion (i.e., urine albumin:creatinine ratio) will be checked prior to enrollment in two separate (collected at least one week apart) spot early morning urine specimens
* Females of child bearing potential must have a negative pregnancy test at screening. Females considered not of childbearing potential include those who have been in menopause at least 2 years, had tubal ligation at least 1 year prior to screening or who have had a total hysterectomy

Exclusion Criteria:

* Use of a BB in the 3 months prior to study enrollment, other than atenolol or metoprolol
* Uncontrolled hypertension with a blood pressure > 160/100 mm Hg or those with changes to their antihypertensive regime during the last 2 months
* Concurrent disease or conditions that would interfere with study participation or safety, such as bleeding disorders, history of syncope or vertigo, severe gastrointestinal reflux (GERD) or gastric ulcers, heart failure, symptomatic coronary or peripheral vascular disease, arrhythmia, serious neurological disorders including seizures or organ transplantation
* Diabetics that are uncontrolled (HbA1c consistently > 9.0 g/dL), unstable, newly diagnosed, or have undergone major changes in therapy within the last 2 months
* Any severe co-morbid condition that would limit life expectancy to < 6 months
* Advanced CKD with an eGFR < 20 ml/min/1.73 m²
* Patients with albuminuria due to causes other than diabetes mellitus or hypertension
* Hepatic enzyme concentrations > 2 times the upper limit of normal
* HIV infection, hepatic cirrhosis or other preexisting liver disease; or positive HIV, Hepatitis B or C test at screening
* Use of any investigational product or investigational medical device within the last 60 days of screening
* History of alcohol and or drug abuse
* Any condition that in view of the investigators places the subject at high risk of poor treatment or compliance or of not completing the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 patients with CKD meeting the inclusion and exclusion criteria listed below will after informed consent be randomized to either nebivolol or sustained release metoprolol succinate and followed for 3 months or early termination of the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy | Baseline to End of Study
  The primary efficacy variable will be the change in ADMA level from baseline to end of study.

SECONDARY OUTCOMES:
Secondary Efficacy | Baseline to End of Study
  Secondary efficacy parameters will include: the change in blood pressure, GFR, urinary albumin excretion, and biomarkers including urinary F2-Isoprostanes, BNP, hsCRP, Cystatin C, and a measure of insulin resistance-the homeostatic model assessment (HOMA) from baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Saran, MD, MS, MRCP, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States